CLINICAL TRIAL: NCT05921214
Title: Identification of Treatment Parameters That Maximize Language Treatment Efficacy For Children
Brief Title: The Effect of Semantic Support on Word Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Late Talker Phase 5; 2R01DC015642-06 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Language Development Disorders
Keywords: Late Talkers
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Using treatment effect sizes, children will be compared to themselves (treatment words v. control words) and across groups (familiar word group v. less-familiar word group).
Who Masked: Participant, Care Provider
Masking Description: The late talkers and their caregivers will not explicitly be told what condition their child is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Familiar Words (Experimental): In this condition, children will learn new words that come from semantic categories (e.g., animals, body parts) from which they currently understand at least several words.
  Interventions: Behavioral: VAULT Phase 5
- Less-Familiar Words (Active Comparator): In this condition, children will learn new words that come from semantic categories (e.g., animals, body parts) from which they currently understand few or no words.
  Interventions: Behavioral: VAULT Phase 5

INTERVENTIONS:
Behavioral: VAULT Phase 5 — This is an input-based vocabulary learning treatment based on principles of statistical learning.

SUMMARY:
The goal of this clinical trial is to compare word learning outcomes in late talking toddlers who are taught different types of words. The main question it aims to answer is if teaching words that come from categories that children already know (e.g., animals) will aid overall word learning. Children will take part in the Vocabulary Acquisition and Usage for Late Talkers (VAULT) word learning treatment and be taught words from more familiar or less familiar categories to see which group learns more words overall.

DETAILED DESCRIPTION:
Children will be assigned to either the familiar or less-familiar word group. All children will receive 8 weeks of Vocabulary Acquisition and Usage for Late Talkers (VAULT) word learning treatment (2x/wk for 30 minutes each session). The investigators will measure how well children learn the words they are taught as well as the words that are in the environment, but not explicitly taught (control words). This will help us know if their learning is due to treatment or maturation. The investigators will compare children to themselves (taught words v. control words) to ensure that the overall treatment is working. Then, the investigators will compare children in the familiar word group to children in the less-familiar word group to see which group learns more overall.

ELIGIBILITY:
Inclusion Criteria:

* Native English Speaking
* Pass pure tone hearing screening or medical report of normal hearing
* 2-3 Years of age
* MCDI expressive scale <10th percentile

Exclusion Criteria:

* Parental report of other diagnoses
* Enrolled in concurrent treatment elsewhere
* Nonverbal IQ <75 as measured by the Bayley scales
* Parents unable to consistently bring child to treatment sessions

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Effect Size | Change from baseline through treatment, which will average an 8-week time frame.
  The investigators will count the number of spontaneous and probed productions of target and control words and calculate a treatment effect size (d).
Number/Rate of Words Learned | Change from Initial Evaluation through Follow-up, which will average a 6-month time frame.
  The investigators will measure the number of words learned and rate of words learned as reported by the parent on the MCDI starting prior to treatment, and measured during, immediately following, and 4-6 weeks after treatment.

SECONDARY OUTCOMES:
Post Treatment Retention | Change from end of treatment to follow up, which will average 4-6 weeks.
  The investigators will use probe data and parental report to determine how many words the child retained from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Alt, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No